CLINICAL TRIAL: NCT05808270
Title: Efficacy of the Application of the Nutrition Care Process on the Eating Habits of Older Adults in the State of Colima During 12 Months of Follow-up: a Randomized, Single-blind Clinical Trial.
Brief Title: Nutrition Care Process in Mexican Older Adults
Acronym: NCP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Colima (Other)
Responsible Party: Principal Investigator, Miguel Huerta, Professor, Universidad de Colima
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Universidad de Colima
Record Dates: First submitted 2023-03-06; First posted 2023-04-11 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Malnutrition
Keywords: Nutrition care process; Older adults; Malnutrition; Eating habits
MeSH Terms: conditions — Malnutrition; Feeding Behavior

STUDY DESIGN:
Intervention Model Description: There will be two groups in which one group will be given a conventional intervention, a second group will use the nutrition care process (NCP). A nutritional clinical history will be applied to each of the older adults to know general data, body composition, biochemical and clinical parameters, nutritional evaluation (considered step 1 of the NCP), then a nutritional diagnosis will be given (step 2) , to give a dietary prescription, objectives, action plan, intervention and nutritional education to the patient for a period of 8 weeks (step 3) to monitor adherence to the nutritional prescription, which will be monitored at 3 , 6 and 12 months (step 4).
Who Masked: Participant
Masking Description: Each participant belonging to this institution has the same probability of being selected for the study. On this occasion, a numbered list of the subjects candidates to participate in the study will be needed. Subsequently, by means of a raffle with balls numbered from 1 to 2, the subjects will be assigned to each of the interventions, number 1 corresponds to the intervention with the nutrition care process and number 2 to the conventional nutritional intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutrition care process (Active Comparator)
  Interventions: Behavioral: Nutrition care process
- Conventional nutritional intervention (Placebo Comparator)
  Interventions: Behavioral: Nutrition care process

INTERVENTIONS:
Behavioral: Nutrition care process — According to the randomization and simple blinding, there will be 2 study groups in which group 1 will be operated on Nutrition care process and group 2 with Conventional nutritional intervention.
  * The Nutrition Care Process is a standardized model intended to guide RDNs in providing high quality nutrition care. The NCP consists of four distinct, interrelated steps: Nutrition Assessment, Diagnosis, Intervention, and Monitoring/Evaluation (AND, 2023).
  * In the case of Conventional nutritional intervention, we will base ourselves on the application of a habitual nutritional clinical history, where information will be obtained on the reasons for consultation and the specific needs of the patient to carry out an intervention based on their priorities.

SUMMARY:
The aim of this clinical trial is to determine the efficacy at 12 months of the application of the nutrition care process in the eating habits of older adults in the state of Colima, Mexico compared to a conventional nutritional intervention.

The main questions it aims to answer is: what is the efficacy of the application of the nutrition care process vs. a conventional nutritional intervention on the eating habits of older adults in the state of Colima, Mexico after 12 months of follow-up?

DETAILED DESCRIPTION:
Participants will be two study groups. Group 1 will apply the nutritional care process and Group 2 will use standard care. The Structured Survey of Food Quality of the older adult will be applied to classify eating habits as good and bad; as well as the reduction of malnutrition in the study participants, in addition, the 24-hour reminder and the food consumption frequency questionnaire will be evaluated before and after the nutritional intervention, an eating plan will be determined according to the needs and later, follow-up will be given for 8 weeks, finally monitoring will be done at 3, 6 and 12 months in order to detect changes in eating habits.

The financial resources will be financed by resources own in the Social Coexistence Center for the older adults in the metropolitan area of Colima, Mexico. Group experience: there are health professionals specialized in patient care.

The protocol has the approval of a local research ethics committee (CEICANCL220223-NUTRICIA-02).

ELIGIBILITY:
Inclusion Criteria:

* Older adults ≥ 60 years old
* female or male
* who voluntarily agree to participate in the study.

Exclusion Criteria:

* People who have a specific treatment determined by another health professional
* people with chronic kidney disease and hemodialysis or dialysis treatment.
* adherence less than 80% in the nutritional intervention
* incomplete data collection, participants who decide to leave the project
* people who are hospitalized or die.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline Eating Habits (Survey of Food Quality of the Older Person) at 12 months | 12 months after the intervention with the Nutrition Care Process
  Application of the structured Survey of Food Quality of the Older Person.
Changes from baseline Malnutrition parameters measured by GLIM Criteria at 12 months | 12 months after the intervention with the Nutrition Care Process
  Application of the Global Leadership Initiative on Malnutrition (GLIM)

SECONDARY OUTCOMES:
Changes from baseline Quality of life perception (WHOQOL) at 12 months | 12 months after the intervention with the Nutrition Care Process
  Application of the Quality of life perception (World Health Organization Quality of Life Questionnaire)
Changes from lean body mass at 12 months | 12 months after the intervention with the Nutrition Care Process
  Lean body mass measured by Bioelectrical Impedance Analysis (Tanita BC 568)
Changes from baseline water mass at 12 months | 12 months after the intervention with the Nutrition Care Process
  Water mass measured by Bioelectrical Impedance Analysis (Tanita BC 568)
Changes from baseline fat body mass at 12 months | 12 months after the intervention with the Nutrition Care Process
  Fat body mass measured by Bioelectrical Impedance Analysis (Tanita BC 568)
Changes from baseline body mass index at 12 months | 12 months after the intervention with the Nutrition Care Process
  weight (Tanita BC 568) and height (SECA 213) will be combined to report BMI in kg/m^2
Changes from baseline energy intake (by a dietary recall) at 12 months | 12 months after the intervention with the Nutrition Care Process
  Calorie intake measured by a 24 food dietary recall and reported in kcal.
Changes from baseline carbohydrate intake (by a dietary recall) at 12 months | 12 months after the intervention with the Nutrition Care Process
  Carbohydrate intake measured by a 24 food dietary recall and reported in grams.
Changes from baseline protein intake (by a dietary recall) at 12 months | 12 months after the intervention with the Nutrition Care Process
  Protein intake measured by a 24 food dietary recall and reported in grams.
Changes from baseline lipid intake (by a dietary recall) at 12 months | 12 months after the intervention with the Nutrition Care Process
  Lipid intake measured by a 24 food dietary recall and reported in grams.
Changes from baseline diabetes mellitus control at 12 months | 12 months after the intervention with the Nutrition Care Process
  diabetes mellitus control reported by a medical record
Changes from baseline obesity control at 12 months | 12 months after the intervention with the Nutrition Care Process
  Obesity control reported by a medical record
Changes from baseline undernutrition control at 12 months | 12 months after the intervention with the Nutrition Care Process
  Undernutrition control reported by a medical record
Changes from baseline hypertension control at 12 months | 12 months after the intervention with the Nutrition Care Process
  Hypertension control reported by a medical record
Changes from baseline serum albumin at 12 months | 12 months after the intervention with the Nutrition Care Process
  Measurement of albumin (g/dL) by serum blood sample (using a Spinreact kit).
Changes from baseline serum total cholesterol at 12 months | 12 months after the intervention with the Nutrition Care Process
  Measurement of total cholesterol (mg/dL) by serum blood sample (using a Spinreact kit).
Changes from baseline serum HDL Cholesterol at 12 months | 12 months after the intervention with the Nutrition Care Process
  Measurement of HDL Cholesterol (mg/dL) by serum blood sample (using a Spinreact kit).
Changes from baseline serum triglycerides at 12 months | 12 months after the intervention with the Nutrition Care Process
  Measurement of triglycerides (mg/dL) by serum blood sample (using a Spinreact kit).
Changes from baseline fasting glucose at 12 months | 12 months after the intervention with the Nutrition Care Process
  Measurement of fasting glucose (mg/dL) by serum blood sample (using a Spinreact kit).

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Huerta, PhD, Study Chair — Universyty of Colima
Locations (1):
- DIF Estatal Colima, Colima, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Academy of Nutrition and Dietetics. Nutrition Care Process — https://www.ncpro.org/nutrition-care-process